CLINICAL TRIAL: NCT04665479
Title: Web-based Digital-storytelling Intervention for Rural-dwelling Children With Life-threatening Conditions
Brief Title: Digital-storytelling Intervention for Rural-dwelling Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Rita & Alex Hillman Foundation (Unknown)
Responsible Party: Principal Investigator, Terrah Akard, Associate Professor, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 123456
Record Dates: First submitted 2020-10-22; First posted 2020-12-11 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Pediatrics
Keywords: Pediatric Palliative Care; Digital Storytelling

STUDY DESIGN:
Intervention Model Description: One group pre- and post-test clinical trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): A total of 30 children with any progressively declining (acute or chronic) life-threatening diagnosis per parent report (aged 8 to 17) and their primary parent caregivers will be recruited as a dyad. Dyads will participate in a nurse-delivered intervention that will guide children to create electronic digital storyboards about themselves during 6 sessions over 6 weeks.
  Interventions: Other: Web-based legacy-making intervention through digital storytelling

INTERVENTIONS:
Other: Web-based legacy-making intervention through digital storytelling — A child-parent dyad will participate in a nurse-delivered intervention that will guide children to create electronic digital storyboards about themselves during 6 sessions over 6 weeks.

SUMMARY:
The overall purpose of this study is to test the feasibility of a web-based storytelling intervention for rural-dwelling children (ages 8-17) with serious advanced illnesses.

There is a growing need for home-based end-of-life and palliative care for children with serious illnesses. While palliative care interventions offered in home settings are significantly lacking, the problems are magnified by substantial gaps in access to palliative care for rural populations. Web-based recruitment and intervention methods have the potential to access hard-to-reach rural populations and provide a cost-effective health care. In particular, legacy-making (i.e., actions/behaviors aimed at being remembered) is one strategy to help decrease suffering and improve psychosocial outcomes for children with serious illness and end of life needs. Storytelling has successfully documented child legacies and may be an ideal format for children. Guided by our existing, web-based digital storytelling intervention and previous work, this project will offer a remotely-delivered legacy-making intervention to rural-dwelling children with diverse serious, advanced health conditions and their parents.

DETAILED DESCRIPTION:
Background: Nearly 1 million children between the ages of 8 and 17 years worldwide are estimated to be in need of palliative care. These children and their parents are at substantial risk for suffering and long-term morbidity. Pediatric palliative care interventions have primarily focused on children with cancer, despite children with cancer only representing 30 to 40% of patients receiving pediatric palliative care services. Despite parents preferring that children with serious illnesses die at home, nearly two-thirds of children die in hospital or care facilities. The need for home-based end-of-life and palliative care is critical for this vulnerable population, yet interventions offered in home settings are significantly lacking. Risks are magnified by substantial gaps in access to palliative care for rural populations. Challenges to care for rural-dwelling children with serious illnesses and their caregivers include lack of pediatric-focused local healthcare resources; need to move residence; disruption to family life; missed school; financial burdens from missed work and costs associated with food, gas, and housing; and a lack of communication between urban and rural healthcare providers. Thus, the burden for children with serious illnesses and their parents may be greater for those living in rural versus urban communities.

Legacy-making (i.e., actions/behaviors aimed at being remembered) is one strategy to help decrease suffering and improve psychosocial outcomes for individuals with serious illness and end of life needs. Storytelling has successfully documented child legacies and may be an ideal format for children. Our interdisciplinary team, rooted in nursing's unique perspective, has successfully developed and tested a digital storytelling intervention in pediatric oncology. Parents reported that the intervention facilitated "conversations with [ill child] that I otherwise wouldn't have had." One parent said, "This project was really a neat way for [ill child] to express himself…. He loved picking out photos and thinking about his favorites…. we worked together, and it really did create a bond." Research in this field has yet to expand outside of oncology or to rural settings, and we have significantly modified our existing digital storytelling intervention based on parent input to further increase its effect. In the proposed project, guided by our conceptual framework based on our previous work and existing theory, our goal is to expand to non-cancer pediatric patients and determine the feasibility of our newly adapted intervention for rural-dwelling children with diverse serious, advanced conditions and their parents.

Objective/Hypothesis: The overall purpose of this study is to test the feasibility of a web-based storytelling intervention for rural-dwelling children (ages 8-17) with serious advanced illnesses.

Specific aims are to: (1) determine feasibility and acceptability of a digital storytelling intervention for rural-dwelling children with serious illness; (2) determine the feasibility of data collection procedures, and (3) determine child and parent perceptions of the benefits of storytelling.

Study Design: One group pre- and post-test clinical trial design will be used. A total of 30 children with any progressively declining (acute or chronic) life-threatening diagnosis per parent report (aged 8 to 17) and their primary parent caregivers will be recruited via Facebook (N=30 dyads; 60 total participants). Dyads will participate in a nurse-delivered intervention that will guide children to create electronic digital storyboards about themselves during 6 sessions over 6 weeks. A trained nurse will deliver sessions averaging 1 hour each via Zoom. Dyads will receive a final digital story that plays in a cinematic format. Participants will be asked to complete baseline and post-intervention measures, attempting to assess following outcome variables: (a) child psychological distress, (b) parent psychological distress, (c) parent-child communication, (d) family relationships, and (e) program satisfaction.

ELIGIBILITY:
Inclusion Criteria for Children:

* any progressively declining (acute or chronic) life-threatening diagnosis per parent report
* living in a rural area based on the Federal Office of Rural Health Policy criteria (https://www.hrsa.gov/rural-health/about-us/definition/datafiles.html)
* speak and understand English

Inclusion Criteria for Parents:

* 18 years of age and older
* child's primary parent caregiver
* speak and understand English
* living in a rural area based on the Federal Office of Rural Health Policy criteria (https://www.hrsa.gov/rural-health/about-us/definition/datafiles.html)

Exclusion Criteria:

* currently live outside of the United States or live in a non-rural area
* have any cognitive impairment(s) per parent report
* do not have internet access and/or electronic devices (e.g., laptop, desktop computer, mobile phone, tablet PC) required for the study participation

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in PROMIS Pediatric Psychological Distress - Short Form | Day 0, Day 43
  A 8-item 5-point Likert scale measure ranging from 1 (never) to 5 (always) to assess children's psychological distress.
Change in PROMIS Pediatric Anxiety - Short Form | Day 0, Day 43
  A 8-item 5-point Likert scale measure ranging from 1 (never) to 5 (almost always) to assess children's anxiety.
Change in PROMIS Pediatric Depressive Symptom - Short Form | Day 0, Day 43
  A 8-item 5-point Likert scale measure ranging from 1 (never) to 5 (almost always) to assess children's depressive symptoms.
Change in PROMIS Pediatric Meaning and Purpose - Short Form | Day 0, Day 43
  A 8-item 5-point Likert scale measure ranging from 1 (not at all) to 5 (very much) to assess children's perception of meaning and purpose of life.
Change in NIH Toolbox Perceived Stress Survey | Day 0, Day 43
  A 10-item 5-point Likert scale measure ranging from 1 (never) to 5 (very often) to assess parents' perceived stress in the past month.
Change in PROMIS Anxiety - Short Form | Day 0, Day 43
  A 8-item 5-point Likert scale measure ranging from 1 (never) to 5 (always) to assess parents' anxiety.
Change in PROMIS Depression- Short Form | Day 0, Day 43
  A 8-item 5-point Likert scale measure ranging from 1 (never) to 5 (always) to assess parents' depression.
Change in PROMIS Meaning and Purpose - Short Form | Day 0, Day 43
  A 8-item 5-point Likert scale measure ranging from 1 (strongly disagree) to 5 (strongly agree) to assess parents' perception of meaning and purpose of life.
Change in Parent-Adolescent Communication Scale | Day 0, Day 43
  A 20-item 5-point Likert scale measure ranging from 1 (strongly disagree) to 5 (strongly agree) to assess quality of parent-adolescent communication.
Change in PROMIS Pediatric Family Relationships - Short Form | Day 0, Day 43
  A 8-item 5-point Likert scale measure ranging from 1 (never) to 5 (always) to assess children's perception of family relationships.
Satisfaction Survey | Day 43
  A 16-item survey to assess participants' satisfaction of the intervention program. Ten 7-point Likert scale items assess satisfaction, and 6 items assess perceived benefits of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Terrah Akard, PhD, Principal Investigator — Vanderbilt University School of Nursing
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
There are no tangible resources to share at this time as the intervention is in testing phases. We plan to make the intervention available for sharing in the future, upon completed testing. Therefore, data is the only resource available for sharing.
  The proposed research will produce data with 30 rural-dwelling children with serious health conditions-parent dyads. The final data set will contain demographic information and children/parent responses on psychological distress, family relationship, and communication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for sharing no later than the publication date of the main results from the final dataset. Data will be disclosed without a specific deadline.
Access Criteria: The data will be shared with anyone who is interested in this study. We especially seek to make our data available to the community of scientists interested in pediatric palliative care, specifically related to rural-dwelling children with life-threatening conditions and their parents.